CLINICAL TRIAL: NCT06413888
Title: Routine Nasogastric Drainage vs. No Drainage Using Nasogastric Tube After Pancreaticoduodenectomy: A Randomized Control Trial [NCT ID Not Yet Assigned]
Brief Title: Nasogastric Decompression Following Pancreaticoduodenectomy
Acronym: whipple
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Omar Barakat, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-43383
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Head Neoplasm; Delayed Gastric Emptying; Post Operative Ileus; Whipple Procedure
MeSH Terms: conditions — Gastroparesis | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Intervention Model Description: Two groups of patients. Group 1 patients will have NGT placed in the operating room and continued in the immediate postoperative recovery period. Group 2 patients will have oropharyngeal gastric tube inserted in the operating room and removed at the end of the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A ( No NGT) (Active Comparator)
  Interventions: Procedure: pancreaticoduodenectomy
- Group B (NGT Retained) (Active Comparator)
  Interventions: Procedure: pancreaticoduodenectomy

INTERVENTIONS:
Procedure: pancreaticoduodenectomy — Surgical removal of the head of the pancreas, duodenum, extrahepatic bile duct, distal stomach, and proximal jejunum. Group A cohort will not have NGT placed in the postoperative period. Whereas, group B will have the NGT retained in the posoperative period
  Other Names: Whipple

SUMMARY:
Pancreaticoduodenectomy (PD) remains the gold-standard operation for peri-ampullary neoplasms. Traditionally, gastric decompression via nasogastric intubation has been employed postoperatively to prevent nausea, vomiting, aspiration pneumonia, anastomotic leakage and delayed gastric emptying. Recently, the implementation of ERAS protocol recommended against routine use of nasogastric tube following PD. however, limited data exists surrounding the identification of those patients needing NGT decompression in the immediate postoperative period. Therefore, we initiated a large prospective randomized controlled trial to evaluate the clinical outcomes of patients who retained the NGT post-PD versus those who had it removed at the end of the procedure. This study aims to assess the effectiveness of nasogastric decompression in PD recovery, with the primary endo point being the need for and impact of NGT in the postoperative recovery. The secondary endpoint will examined the re-insertion rate of NGT and identify factors that necessitate its use in the immediate postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older
* Patients undergoing successful pancreaticoduodenectomy for benign or malignant neoplasm.

Exclusion Criteria:

* Patients who does not complete the procedure due to locally advanced or metastatic disease discovered during the procedure.
* Patient who requires prolong postoperative intubation in the postoperative period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
to assess whether nasogastric decompression following a whipple procedure will reduce the incidence and severity of postoperative complications | 30-days postoperatively
  Severity of post operative complications was graded according to the Clavien-Dindo classification system adopted for pancreaic surgery, which relies on the type of treatment used for each complication with scores range from 1-4, and any complication graded >2 considered a major complication.

SECONDARY OUTCOMES:
Examined the re-insertion rate of Nasogastric tube following pancreaticoduodenectomy | 30- days postoperatively
  Patient will be considered to undergo nasogastric decompression with nasogastric tube if he/she demonstrated clinical evidence of postoperative ileus and delayed gastric emptying as defined according to the consensus definition proposed by the international study group of pancreatic surgery (ISGPS), the severity of which was classified into 3 grades (A,B, and C) based on clinical course and postoperative management such as the need nausea and vomiting and inability to tolerate solid oral intake by the end of the first postoperative week.
identify factors that necessitated its use in the immediate postoperative period | 30 days postoperatively
  To identify preoperative factors such as obesity with BMI 30 or more, Preoperative uncontrolled diabtes, older age (over 70), gender (male/female), histroy of gastric outlet obstruction, primary diagnosis (malignant disease vs benign). Intra-operative factor such such as the length of the procedure, blood loss, any concurrent procedure such as extensive lysis of adhesions, colon resection; and postoperative factors including postoperative blood counts, phosphorus and magnesium levels, blood sugar level, and postoperative complications. These factors will be assessed using logistic regression analysis to predict the necessity of nasogastric decompression in the postoperative period following the whipple procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Barakat, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor college of medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No